CLINICAL TRIAL: NCT03881059
Title: A Randomized, Placebo-Controlled, Double-blind, Multicenter Study to Assess the Efficacy and Safety of Multiple Doses of BMS-986165 in Subjects With Active Psoriatic Arthritis (PsA)
Brief Title: Efficacy and Safety of BMS-986165 Compared With Placebo in Participants With Active Psoriatic Arthritis (PsA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-084; 2018-004293-10 (EudraCT Number)
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Active Psoriatic Arthritis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigative site staff, the Sponsor, and Participant will remain blinded to treatment assignment with the exception of an unblinded pharmacist, an unblinded study drug administrator (Part B), and an unblinded site monitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Placebo (Placebo Comparator)
  Interventions: Other: BMS-986165 Placebo
- Part A: BMS-986165 Dose A (Experimental)
  Interventions: Drug: BMS-986165 Dose A
- Part A: BMS-986165 Dose B (Experimental)
  Interventions: Drug: BMS-986165 Dose B
- Part B: Ustekinumab + BMS-986165 Placebo (Experimental)
  Interventions: Other: BMS-986165 Placebo; Drug: Ustekinumab
- Part B: BMS-986165 Dose A + Ustekinumab Placebo (Experimental)
  Interventions: Drug: BMS-986165 Dose A; Other: Ustekinumab Placebo
- Part B: BMS-986165 Dose B + Ustekinumab Placebo (Experimental)
  Interventions: Drug: BMS-986165 Dose B; Other: Ustekinumab Placebo

INTERVENTIONS:
Other: BMS-986165 Placebo — Participants will receive BMS-986165 matching placebo QD
  Arms: Part A: Placebo; Part B: Ustekinumab + BMS-986165 Placebo
Drug: BMS-986165 Dose A — Participants will receive BMS-986165 Dose A QD.
  Arms: Part A: BMS-986165 Dose A; Part B: BMS-986165 Dose A + Ustekinumab Placebo
Drug: BMS-986165 Dose B — Participants will receive BMS-986165 dose B QD.
  Arms: Part A: BMS-986165 Dose B; Part B: BMS-986165 Dose B + Ustekinumab Placebo
Drug: Ustekinumab — Participants will receive ustekinumab SQ injection QD.
  Arms: Part B: Ustekinumab + BMS-986165 Placebo
Other: Ustekinumab Placebo — Participants will receive ustekinumab SQ matching placebo QD
  Arms: Part B: BMS-986165 Dose A + Ustekinumab Placebo; Part B: BMS-986165 Dose B + Ustekinumab Placebo

SUMMARY:
The main purpose of study is to assess the dose-response relationship of BMS-986165 (Dose A or Dose B once daily [QD]) at Week 16 in the treatment of participants with active PsA.

DETAILED DESCRIPTION:
The study is intended to evaluate the safety and efficacy of BMS-986165 Dose A or B once daily (QD) compared with placebo in adults with active PsA. The primary endpoint is american college of rheumatology (ACR) 20 response at Week 16 (Part A).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PsA for at least 6 months before screening, and who meet the Classification Criteria for Psoriatic Arthritis (CASPAR) at screening
* Participants either (i) cannot have prior exposure to biologics (biologic-naïve) or (ii) have failed or been intolerant to 1 tumor necrosis factor -inhibitor (TNFi) (TNFi-experienced). Failure is defined as lack of response or loss of response with at least 3 months of therapy with an approved dose of a TNFi, as judged by the investigator. Failure must have occurred at least 2 months prior to Day 1
* Participants have at least 1 confirmed greater than or equal to (>=) 2 centimeter (cm) lesion of plaque psoriasis at screening
* Participants have active arthritis as shown by a minimum of >= 3 swollen joints and >= 3 tender joints (66/68 joint counts) at screening and Day 1
* High sensitivity C-reactive protein (hsCRP) >= 3milligram per liter (mg/L) at screening
* Women of Childbearing Potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study treatment

Exclusion Criteria:

* Has non-plaque psoriasis (that is (i.e.), guttate, inverse, pustular, erythrodermic or drug-induced psoriasis) at screening or Day 1
* Has any other autoimmune condition such as rheumatoid arthritis, etc. There are exceptions for inflammatory bowel disease or uveitis as follows: currently active disease is excluded but, a history of no longer active disease for at least 12 months (including not being on medication) is allowed
* Has active (i.e. currently symptomatic) fibromyalgia
* History or evidence of active infection and/or febrile illness within 7 days prior to Day 1 (example, bronchopulmonary, urinary, gastrointestinal, etc.)
* History of recent serious bacterial, fungal, or viral infections requiring hospitalization and intravenous (IV) antimicrobial treatment within 90 days prior to screening, or any infection requiring antimicrobial treatment within 15 days prior to Day 1
* History of active tuberculosis (TB) prior to screening visit, regardless of completion of adequate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (94):
- United States (31):
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Medvin Clinical Research - Covina Office, Covina, California
  - University of California at San Diego Medical Center, La Jolla, California
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Omega Research Consultants - Metrowest, Orlando, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - BayCare Medical Group, St. Petersburg, Florida
  - University of South Florida - Morsani College of Medicine, Tampa, Florida
  - Heartland Research Associates - East Wichita, Wichita, Kansas
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Arthritis Associates, Hattiesburg, Mississippi
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Coast Rheumatology, Toms River, New Jersey
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - The Center for Rheumatology-Albany, Albany, New York
  - University of Rochester Medical Center, Rochester, New York
  - Joint Muscle Medical Care and Research Institute - Lilington Office, Charlotte, North Carolina
  - DJL Clinical Research, Charlotte, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Paramount Medical Research and Consulting, Middleburg Heights, Ohio
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Office of Ramesh C. Gupta, MD, Memphis, Tennessee
  - Pioneer Research Solutions, Cypress, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
- Czechia (9):
  - L.K.N. Arthrocentrum, s.r.o, Hlu?
  - CCR Ostrava, Ostrava
  - Revmatologie MUDr. Klara Sirova s.r.o., Ostrava
  - Arthrocentrum, Prague
  - Revmatologicky Ustav, Prague
  - CCR Prague, Prague
  - Nuselska Poliklinika, Prague
  - Affidea Praha, Praha 11 Chodov
  - PV-Medical Services, s.r.o., Zlín
- Germany (8):
  - Charite Universitatsmedizin Berlin, Berlin
  - Rheumatologische Schwerpunktpraxis PD Dr. med. Brandt Jurgens, Berlin
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - HRF II - Hamburger Rheuma Forschungszentrum II - MVZ fur Rheumatologie und Autoimmunmedizin Hamburg, Hamburg
  - SMO.MD GmbH, Magdeburg
  - Universitatsmedizin Mannheim, Mannheim
  - Klinikum der Universitat Munchen, München
- Hungary (7):
  - Clinexpert Gyogycentrum, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Egeszsegugyi es Szolgaltato Korlatolt Felelossegu Tarsasag, Miskolc
  - Aranyklinika, Szeged
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - CMed Rehabilitacios es Diagnosztikai Kozpont, Székesfehérvár
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy
- Poland (20):
  - Osteo-Medic, Bia?ystok
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - ClinicMed Daniluk Nowak Spolka Jawna, Bialystok
  - Nasz Lekarz Osrodek Badan Klinicznych - Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki Number 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Indywidualna Specjalistyczna Praktyka Lekarska Lek. Med. Barbara Bazela, Elblag
  - Malopolskie Badania Kliniczne, Krakow
  - Grazyna Pulka Specjalistyczny Osrodek All-med, Krak
  - Pratia MCM Krakow, Krak
  - AMED Centrum Medyczne, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej Lecznica Mak-Med Spolka Cywilna, Nadarzyn
  - Centrum Badan Klinicznych S.C., Poznan
  - Ai Centrum Medyczne, Poznan
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Ars Rheumatica - Reumatika Centrum Reumatologii, Warsaw
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw
  - WroMedica, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Russia (10):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Scientific Research Medical Complex, Kazan'
  - Medical Center Revma-Med, Kemerovo
  - Clinic on Maroseyka, Moscow
  - Medical Center Health Family, Novosibirsk
  - State Healthcare Institution of the Republic of Karelia-Republican Hospital im.V.A.Baranova, Petrozavodsk
  - Clinical Rheumatological Hospital Number 25, Saint Petersburg
  - Polyclinic of Private Security Personnel, Saint Petersburg
  - LLC Medical Consultation and Research Center-Practice, Yarolavl
  - Clinical Hospital named after NA Semashko, Yaroslavl
- Spain (6):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - The Princess Alexandra Hospital NHS Trust, Harlow

REFERENCES:
- [Derived] Deodhar A, Nowak M, Ye JY, Lehman T, Banerjee S, Mease PJ. Efficacy and Safety of Deucravacitinib, a Selective, Allosteric TYK2 Inhibitor, by Baseline DMARD Use in a Phase 2 Psoriatic Arthritis Study: A Post Hoc Analysis. Rheumatol Ther. 2025 Oct;12(5):873-887. doi: 10.1007/s40744-025-00776-4. Epub 2025 Jul 5. PMID 40616721
- [Derived] FitzGerald O, Gladman DD, Mease PJ, Ritchlin C, Smolen JS, Gao L, Hu Y, Nowak M, Banerjee S, Catlett I. Phase 2 Trial of Deucravacitinib in Psoriatic Arthritis: Biomarkers Associated With Disease Activity, Pharmacodynamics, and Clinical Responses. Arthritis Rheumatol. 2024 Sep;76(9):1397-1407. doi: 10.1002/art.42921. Epub 2024 Jul 1. PMID 38770592
- [Derived] Strand V, Gossec L, Coates LC, Ogdie A, Choi J, Becker B, Zhuo J, Lehman T, Nowak M, Elegbe A, Mease PJ, Deodhar A. Improvements in Patient-Reported Outcomes After Treatment With Deucravacitinib in Patients With Psoriatic Arthritis: Results From a Randomized Phase 2 Trial. Arthritis Care Res (Hoboken). 2024 Aug;76(8):1139-1148. doi: 10.1002/acr.25333. Epub 2024 May 7. PMID 38529674
- [Derived] Mease PJ, Deodhar AA, van der Heijde D, Behrens F, Kivitz AJ, Neal J, Kim J, Singhal S, Nowak M, Banerjee S. Efficacy and safety of selective TYK2 inhibitor, deucravacitinib, in a phase II trial in psoriatic arthritis. Ann Rheum Dis. 2022 Jun;81(6):815-822. doi: 10.1136/annrheumdis-2021-221664. Epub 2022 Mar 3. PMID 35241426
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 203 participants were randomized and treated.
Groups:
- Placebo: In Part A, Placebo matching BMS-986165. In Part B, Ustekinumab SQ.
- BMS-986165 6 mg: In Part A, BMS-986165 6 mg administered QD for 16 weeks. In Part B, participants received either BMS-986165 at 6 mg (if they achieved minimal disease activity (MDA) in Part A) or Ustekinumab SQ (if they did not achieve MDA in Part A)
- BMS-986165 12 mg: In Part A, BMS-986165 12 mg administered QD for 16 weeks. In Part B, participants received either BMS-986165 at 12 mg (if they achieved minimal disease activity (MDA) in Part A) or Ustekinumab SQ (if they did not achieve MDA in Part A)
Period: Treatment Period - Part A
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Started | 66 | 70 | 67
Completed | 58 | 63 | 59
Not Completed | 8 | 7 | 8
Not completed — Adverse Event | 1 | 3 | 4
Not completed — Randomized by mistake with study treatment | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 3
Not completed — Other reasons | 2 | 1 | 0
Period: Treatment Period - Part B
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Started (Participation in Part B was optional. Some of the participants who completed Part A decided not to continue in Part B) | 55 | 60 | 58
Participants Maintaining Same Treatment as in Part A | 0 | 13 | 16
Participants Treated With Ustekinumab in Part B | 55 | 47 | 42
Completed | 47 | 54 | 47
Not Completed | 8 | 6 | 11
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Death | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Site terminated by sponsor | 1 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Other reasons | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg | Total
Number analyzed (Participants) | 66 | 70 | 67 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (13.17) | 50.5 (13.69) | 50.5 (13.75) | 49.8 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 30 | 34 | 104
  Male | 26 | 40 | 33 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 5 | 16
  Not Hispanic or Latino | 59 | 65 | 62 | 186
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 65 | 67 | 67 | 199
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving the American College of Rheumatology (ACR) 20 Response at Week 16
Description: A participant is considered an ACR 20 responder if the following three conditions are met: 1) ≥ 20% improvement from baseline in the number of tender joints (68 joint count). 2) ≥ 20% improvement from baseline in the number of swollen joints (66 joint count). 3) ≥ 20% improvement from baseline in at least 3 of the following 5 domains: o Subject Global Assessment of disease activity o Physician Global Assessment of psoriatic arthritis o Subject Global Assessment of pain o Health Assessment Questionnaire-Disability Index (HAQ-DI) o High-sensitivity C-reactive protein (hsCRP)
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 31.8 [20.6 to 43.1] | 52.9 [41.2 to 64.6] | 62.7 [51.1 to 74.3]
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 6 mg vs BMS-986165 12 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Slope Coefficient of Dose = 0.11, 95% CI 2-sided [0.05 to 0.17]

2. Secondary Outcome: Adjusted Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI is measured by the use of a patient-reported outcome measure questionnaire, assessing the degree of difficulty a person has experienced during the past week in 8 domains of daily living activities. Each activity category consists of 2 to 3 questions (total of 20 questions). For reach question the level of activity is scored from 0 to 3, with 0 representing "no difficulty" and 3 as "unable to do". Any activity that requires assistance from another individual or an assistive device adjusts to a minimum score of 2. For each activity category, the highest score reported in the 2 or 3 questions pertinent to that category represents the category score. Scores from the 8 categories are then summed and divided by 8 to generate the final score. The final score can range from 0 (most desirable outcome) to 3 (least desirable outcome). Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | -0.11 (0.066) | -0.37 (0.065) | -0.39 (0.067)

3. Secondary Outcome: Percentage of Participants Achieving the Psoriasis Area and Severity Index (PASI) 75 Response
Description: The PASI is a measure of the average erythema, induration thickness and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI 75 response rate represents the percentage of participants who experienced at least a 75% improvement in PASI score as compared with the baseline value. PASI assessment was performed by trained professionals.
Time Frame: 16 weeks after first dose
Population: All treated participants with at least 3% Body Surface Area (BSA) involvement at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 54 | 59 | 52
Percent of Participants | 20.4 [9.6 to 31.1] | 42.4 [29.8 to 55.0] | 59.6 [46.3 to 73.0]

4. Secondary Outcome: Adjusted Change From Baseline in the Physical Component Summary (PCS) Score of the Short Form Health Survey-36 (SF-36) Questionnaire
Description: The SF-36 is a patient-reported outcome measure, which includes 36 items in a Likert-type format to measure the following 8 health dimensions over the past week: 1) limitations in physical activities, such as bathing or dressing 2) limitations in social activities because of physical or emotional problems 3) limitations in usual role activities because of physical health problems 4) bodily pain 5) general mental health (psychological distress and well-being) 6) limitations in usual role activities because of emotional problems 7) vitality (energy and fatigue) and 8) general health perceptions. The 8 health dimensions assessed are grouped into 2 main components, physical and mental. Each of the 8 dimensions contribute to both the Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score. PCS and MCS scores range from 0 to 100, with high scores indicating a better health status. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | 2.3 (0.97) | 5.6 (0.94) | 5.8 (0.97)

5. Secondary Outcome: Percentage of Participants Achieving the American College of Rheumatology (ACR) 50 Response at Week 16
Description: A participant is considered an ACR 50 responder if the following three conditions are met: 1) ≥ 50% improvement from baseline in the number of tender joints (68 joint count). 2) ≥ 50% improvement from baseline in the number of swollen joints (66 joint count). 3) ≥ 50% improvement from baseline in at least 3 of the following 5 domains: o Subject Global Assessment of disease activity o Physician Global Assessment of psoriatic arthritis o Subject Global Assessment of pain o Health Assessment Questionnaire-Disability Index (HAQ-DI) o High-sensitivity C-reactive protein (hsCRP)
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 10.6 [3.2 to 18.0] | 24.3 [14.2 to 34.3] | 32.8 [21.6 to 44.1]

6. Secondary Outcome: Percentage of Participants Achieving the American College of Rheumatology (ACR) 70 Response at Week 16
Description: A participant is considered an ACR 70 responder if the following three conditions are met: 1) ≥ 70% improvement from baseline in the number of tender joints (68 joint count). 2) ≥ 70% improvement from baseline in the number of swollen joints (66 joint count). 3) ≥ 70% improvement from baseline in at least 3 of the following 5 domains: o Subject Global Assessment of disease activity o Physician Global Assessment of psoriatic arthritis o Subject Global Assessment of pain o Health Assessment Questionnaire-Disability Index (HAQ-DI) o High-sensitivity C-reactive protein (hsCRP)
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 1.5 [0.0 to 4.5] | 14.3 [6.1 to 22.5] | 19.4 [9.9 to 28.9]

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity According to the Disease Activity Score-28 Using C Reactive Protein (DAS 28 CRP)
Description: A Disease Activity Score (DAS) is a scoring system used to assess disease activity. DAS 28 CRP is a composite outcome measure that assesses: • How many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints, but excluding distal interphalangeal joints), wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28. • C Reactive Protein (CRP) levels in the blood (as a measure of the degree of inflammation) • Subject Global Assessment of disease activity The results are combined to produce the DAS 28 CRP score, which correlates with the extent of disease activity as follows: • < 2.6: Disease remission • 2.6 - 3.2: Low disease activity • 3.2 - 5.1: Moderate disease activity • > 5.1: High disease activity. Only participants with a score < 3.2 are considered to have achieved low disease activity.
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 22.7 [12.6 to 32.8] | 37.1 [25.8 to 48.5] | 43.3 [31.4 to 55.1]

8. Secondary Outcome: Percentage of Participants Achieving Remission According to the Disease Activity Score-28 Using C Reactive Protein (DAS 28 CRP)
Description: A Disease Activity Score (DAS) is a scoring system used to assess disease activity. DAS 28 CRP is a composite outcome measure that assesses: • How many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints, but excluding distal interphalangeal joints), wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28. • C Reactive Protein (CRP) levels in the blood (as a measure of the degree of inflammation) • Subject Global Assessment of disease activity The results are combined to produce the DAS 28 CRP score, which correlates with the extent of disease activity as follows: • < 2.6: Disease remission • 2.6 - 3.2: Low disease activity • 3.2 - 5.1: Moderate disease activity • > 5.1: High disease activity. Only participants with a score < 2.6 are considered to have achieved remission.
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 6.1 [0.3 to 11.8] | 24.3 [14.2 to 34.3] | 25.4 [15.0 to 35.8]

9. Secondary Outcome: Adjusted Change From Baseline in the Disease Activity Score-28 Using C Reactive Protein (DAS 28 CRP) Score
Description: A Disease Activity Score (DAS) is a scoring system used to assess disease activity. DAS 28 CRP is a composite outcome measure that assesses: • How many joints in the hands (including metacarpophalangeal and proximal interphalangeal joints, but excluding distal interphalangeal joints), wrists, elbows, shoulders, and knees are swollen and/or tender over a total of 28. • C Reactive Protein (CRP) levels in the blood (as a measure of the degree of inflammation) • Subject Global Assessment of disease activity The results are combined to produce the DAS 28 CRP score, which correlates with the extent of disease activity as follows: • < 2.6: Disease remission • 2.6 - 3.2: Low disease activity • 3.2 - 5.1: Moderate disease activity • > 5.1: High disease activity. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | -0.9 (0.15) | -1.7 (0.15) | -1.7 (0.15)

10. Secondary Outcome: Adjusted Change From Baseline in Dactylitis Count
Description: The number of digits in hands and feet with dactylitis (Tender + Non-Tender) was counted and change from baseline at week 16 was assessed. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with dactylitis count ≥ 1 at baseline
Measure: Mean (Standard Error); unit: Digits with dactylitis
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 25 | 33 | 27
Digits with dactylitis | -1.8 (0.40) | -2.0 (0.38) | -2.5 (0.38)

11. Secondary Outcome: Adjusted Change From Baseline in the Leeds Dactylitis Index (LDI) Basic Score
Description: The Leeds Dactylitis Index (LDI) Basic is a quantitative measurement of dactylitis in the 20 digits using a dactylometer. The circumference of the affected and contralateral digits, and tenderness of the affected digits are measured to generate a total score. For each dactylitic digit, the final score is defined as: [{(A/B) - 1}*100]*C, where A is circumference of involved digit, B is circumference of the opposite, unaffected, digit or reference, and C is tenderness (0 or 1). The total score is determined by summing the relative score of all digits. A higher score indicates worse dactylitis. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with LDI score > 0 at baseline
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 24 | 30 | 23
Score on a scale | -28.3 (8.87) | -41.8 (8.35) | -44.5 (8.90)

12. Secondary Outcome: Percentage of Participants Achieving Dactylitis Resolution
Description: Dactylitis resolution (tender digits only) is defined as a dactylitis count of 0 in participants with dactylitis count ≥ 1 at baseline
Time Frame: 16 weeks after first dose
Population: All treated participants with dactylitis count (tender digits only) ≥ 1 at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 25 | 30 | 24
Percent of Participants | 60.0 [40.8 to 79.2] | 76.7 [61.5 to 91.8] | 79.2 [62.9 to 95.4]

13. Secondary Outcome: Adjusted Change From Baseline in Enthesitis by the Leeds Enthesitis Index (LEI)
Description: The LEI was developed specifically for psoriatic arthritis. An overall score of 0 to 6 is derived from the presence or absence of tenderness at 6 entheseal sites (right and left: lateral epicondyle, medial femoral condyle, and Achilles tendon insertion) at the time of evaluation. A higher count indicates a greater enthesitis burden. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with LEI score ≥ 1 at baseline
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 31 | 39 | 26
Score on a scale | -1.2 (0.27) | -1.5 (0.25) | -1.7 (0.28)

14. Secondary Outcome: Adjusted Change From Baseline in Enthesitis by the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index
Description: The SPARCC Enthesitis Index has a 0 to 16 score that is derived from the evaluation of 8 locations: the greater trochanter (R/L), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial and lateral epicondyles (R/L), and the supraspinatus insertion (R/L). A higher count indicates a higher enthesitis burden based on the current evaluation. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with SPARCC enthesitis index score ≥ 1 at baseline
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 34 | 43 | 34
Score on a scale | -1.2 (0.54) | -2.9 (0.48) | -3.1 (0.51)

15. Secondary Outcome: Percentage of Participants Achieving Enthesitis Resolution by the Leeds Enthesitis Index (LEI)
Description: The LEI was developed specifically for psoriatic arthritis. An overall score of 0 to 6 is derived from the presence or absence of tenderness at 6 entheseal sites (right and left: lateral epicondyle, medial femoral condyle, and Achilles tendon insertion) at the time of evaluation. A higher count indicates a greater enthesitis burden. Enthesitis resolution is defined as s LEI score of 0, in subjects with LEI ≥ 1 at baseline
Time Frame: 16 weeks after first dose
Population: All treated participants with LEI score ≥ 1 at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 31 | 39 | 26
Percent of Participants | 22.6 [7.9 to 37.3] | 51.3 [35.6 to 67.0] | 50.0 [30.8 to 69.2]

16. Secondary Outcome: Percentage of Participants Achieving Enthesitis Resolution by the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index
Description: The SPARCC Enthesitis Index has a 0 to 16 score that is derived from the evaluation of 8 locations: the greater trochanter (R/L), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial and lateral epicondyles (R/L), and the supraspinatus insertion (R/L). A higher count indicates a higher enthesitis burden based on the current evaluation. Enthesitis resolution defined as a SPARCC enthesitis index score of 0, in subjects with SPARCC ≥ 1 at baseline.
Time Frame: 16 weeks after first dose
Population: All treated participants with SPARCC enthesitis index score ≥ 1 at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 34 | 43 | 34
Percent of Participants | 17.6 [4.8 to 30.5] | 51.2 [36.2 to 66.1] | 41.2 [24.6 to 57.7]

17. Secondary Outcome: Percentage of Participants Achieving a Physicians Global Assessment-Fingernails (PGA-F) Score of 0 or 1
Description: In participants with psoriasis fingernail involvement, the PGA-F score is used to evaluate the overall condition of the fingernails in terms of disease severity. The assessment is performed by the investigator, who rates the fingernail condition on a 5-point scale based on the higher of the nail bed/nail matrix score. Scores are 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe).
Time Frame: 16 weeks after first dose
Population: All treated participants with PGA-F score ≥ 3 at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 12 | 14 | 20
Percent of Participants | 0 [0.0 to 0.0] | 21.4 [0.0 to 42.9] | 50.0 [28.1 to 71.9]

18. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) Response
Description: A Minimal Disease Activity (MDA) responder is defined as a participant fulfilling 5 of the following 7 outcomes: • Tender joint count ≤ 1 • Swollen joint count ≤ 1 • Psoriasis Area and Severity Index (PASI) ≤ 1 or body surface area (BSA) ≤ 3% • Subject Global Assessment of pain ≤ 15 • Subject Global Assessment of disease activity ≤ 20 • Health Assessment Questionnaire-Disability Index (HAQ-DI) ≤ 0.5 • Tender entheseal points ≤ 1
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 7.6 [1.2 to 14.0] | 22.9 [13.0 to 32.7] | 23.9 [13.7 to 34.1]

19. Secondary Outcome: Adjusted Change From Baseline in the Psoriatic Arthritis Disease Activity Score (PASDAS)
Description: PASDAS is a composite measure calculated from the Physician Global Assessment of psoriatic arthritis, the Subject Global Assessment of disease activity, the Short Form Health Survey-36 Item (SF-36) Physical Component Summary (PCS), the swollen joint count, the tender joint count, the Leeds Enthesitis Index (LEI), the Leeds Dactylitis Index (LDI) (Basic), and the the levels of high-sensitivity C-reactive Protein (hsCRP). Each item contributes differently to the final score, which ranges from 0 to 10 (higher scores represent a higher level of disease activity). Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 63 | 70 | 66
Score on a scale | -1.1 (0.21) | -2.0 (0.20) | -2.1 (0.20)

20. Secondary Outcome: Adjusted Change From Baseline in the Disease Activity Index for Psoriatic Arthritis Score (DAPSA)
Description: DAPSA is a composite measure to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender/painful joint count 68, swollen joint count 66, Subject Global Assessment of disease activity, Subject Global Assessment of pain, and the levels of C-reactive Protein (CRP). Final scores are interpreted as follows: - ≤4 = Remission (REM) - > 4 and ≤ 28 = moderate disease activity (MDA) - >28 = high disease activity (HDA). Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | -13.3 (2.20) | -23.2 (2.16) | -25.6 (2.23)

21. Secondary Outcome: Percentage of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC)
Description: PsARC consists of 4 measurements: tender/painful joint count, swollen joint count, Physician Global Assessment of psoriatic arthritis, and Subject Global Assessment of pain ≤ 15. In order to be classified as a PsARC responder, participants must achieve improvement in 2 of 4 measures, one of which must be joint pain or swelling, without worsening in any measure.
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 54.5 [42.5 to 66.6] | 75.7 [65.7 to 85.8] | 74.6 [64.2 to 85.0]

22. Secondary Outcome: Adjusted Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: In participants with baseline evidence of Psoriatic Arthritis Spondylitis, symptoms are evaluated using the BASDAI, which consists of a 0 to 100 scale measuring discomfort, pain, and fatigue in response to 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: • Fatigue (medical) • Spinal pain • Joint pain and swelling • Areas of localized tenderness • Morning stiffness duration • Morning stiffness severity A higher count indicates worse disease. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with evidence of psoriatic arthritis spondylitis at baseline
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 15 | 19 | 16
Score on a scale | -1.7 (0.55) | -2.0 (0.48) | -2.2 (0.57)

23. Secondary Outcome: Adjusted Change From Baseline in the Mental Component Summary (MCS) Score of the Short Form Health Survey-36 (SF-36) Questionnaire
Description: as for outcome 4
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | 0.7 (1.00) | 3.6 (0.97) | 3.5 (1.01)

24. Secondary Outcome: Adjusted Change From Baseline in the Psoriatic Arthritis Impact of Disease (PsAID) 12 Score
Description: PsAID is a 12-item self-report that measures psoriatic arthritis symptoms and impact of disease. Each item is scored on a 0 to 10 numeric rating scale, and each item contributes differently to the final score. Weighted scores for each item are summed and divided by 20 to generate the final score, ranging from 0 to 10 (higher values indicate worse health). Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | -1.0 (0.26) | -2.1 (0.26) | -2.3 (0.26)

25. Secondary Outcome: Adjusted Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score
Description: The FACIT-Fatigue instrument is a questionnaire used to evaluate a range of self-reported symptoms over the past week, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The questionnaire is composed of 13 questions (Short Form 13a) and each question is scored from 1 to 5. The final score results from the sum of the scores of the 13 questions, and ranges from 13 (most desirable outcome) to 65 (least desirable outcome). Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 65 | 67 | 65
Score on a scale | 2.8 (1.17) | 5.6 (1.16) | 7.2 (1.18)

26. Secondary Outcome: Adjusted Change From Baseline in the Work Limitation Questionnaire (WLQ) Score
Description: The Work Limitation Questionnaire (WLQ) is a 25-item self-report that measures the on-the-job impact of chronic health conditions and treatment over the past 2 weeks. It focuses on assessing limitations while performing specific job demands from the following 4 domains: 1) Time management: difficulty with handling time and scheduling demands (5 items) 2) Physical demands: ability to perform job tasks that involve bodily strength, movement, endurance, coordination, and flexibility (6 items) 3) Mental-interpersonal demands: cognitively demanding tasks and on-the-job social interactions (9 items) 4) Output demands: concerns reduced work productivity (5 items). Final score ranges from 0 (limited none of the time) to 100 (limited all of the time). The score can be used to calculate a percent of lost work productivity due to a particular disease state. Adjusted change represents a change from baseline based on statistical model.
Time Frame: From baseline (day of the first dose) to 16 weeks after first dose
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Score on a scale | -1.2 (0.69) | -1.9 (0.67) | -2.7 (0.70)

27. Secondary Outcome: Percentage of Participants Achieving Health Assessment Questionnaire-Disability Index (HAQ-DI) 0.35 Response
Description: The HAQ-DI is measured by the use of a patient-reported outcome measure questionnaire, assessing the degree of difficulty a person has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 questions (total of 20 questions). For reach question the level of activity is scored from 0 ("no difficulty") to 3 ("unable to do"). For each activity category, the highest score reported in the 2 or 3 questions pertinent to that category represents the category score. Scores from the 8 categories are then summed and divided by 8 to generate the final score. The final score can range from 0 (most desirable outcome) to 3 (least desirable outcome). A HAQ-DI 0.35 responder is defined as a participant with an improvement from baseline in HAQ-DI score of at least 0.35.
Time Frame: 16 weeks after first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
Percent of Participants | 15.2 [6.5 to 23.8] | 38.6 [27.2 to 50.0] | 40.3 [28.6 to 52.0]

28. Secondary Outcome: Percentage of Participants Achieving the Psoriasis Area and Severity Index (PASI) 90 Response
Description: The PASI is a measure of the average erythema, induration thickness and scaling of psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI 90 response rate represents the percentage of participants who experienced at least a 90% improvement in PASI score as compared with the baseline value. PASI assessment was performed by trained professionals.
Time Frame: 16 weeks after first dose
Population: All treated participants with at least 3% Body Surface Area (BSA) involvement at baseline
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 54 | 59 | 52
Percent of Participants | 9.3 [1.5 to 17.0] | 20.3 [10.1 to 30.6] | 34.6 [21.7 to 47.5]

29. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Results
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 70 | 67
msec
  PR Interval, Aggregate: number analyzed (Participants) | 57 | 63 | 59
  PR Interval, Aggregate | 3.9 (16.40) | 3.2 (17.83) | -2.9 (37.09)
  QRS Duration, Aggregate: number analyzed (Participants) | 57 | 63 | 59
  QRS Duration, Aggregate | -0.5 (9.07) | 3.9 (11.58) | -1.1 (13.55)
  QT Interval, Aggregate: number analyzed (Participants) | 57 | 63 | 59
  QT Interval, Aggregate | 1.4 (27.47) | 2.7 (28.56) | 1.5 (26.81)
  QTcB Interval, Aggregate: number analyzed (Participants) | 23 | 24 | 27
  QTcB Interval, Aggregate | 2.8 (41.79) | -6.7 (24.46) | 0.4 (20.34)
  QTcF Interval, Aggregate: number analyzed (Participants) | 30 | 28 | 21
  QTcF Interval, Aggregate | -0.6 (29.83) | 2.4 (29.62) | 4.4 (22.96)

30. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Heart Rate
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 57 | 63 | 59
beats/min | -0.7 (8.28) | -1.0 (9.84) | 0.0 (8.82)

31. Secondary Outcome: Change From Baseline in Vital Signs - Diastolic Blood Pressure
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 59 | 64 | 60
mmHg | 1.1 (8.67) | -0.9 (6.10) | -1.7 (7.06)

32. Secondary Outcome: Change From Baseline in Vital Signs - Heart Rate
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 59 | 64 | 60
beats/min | 0.7 (9.40) | -2.5 (9.02) | 0.8 (8.56)

33. Secondary Outcome: Change From Baseline in Vital Signs - Respiratory Rate
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 59 | 64 | 60
breaths/min | 0.0 (1.88) | -0.2 (1.46) | 0.2 (1.16)

34. Secondary Outcome: Change From Baseline in Vital Signs - Systolic Blood Pressure
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 59 | 64 | 60
mmHg | 1.6 (11.05) | -0.6 (10.95) | -1.5 (11.44)

35. Secondary Outcome: Change From Baseline in Vital Signs - Temperature
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: Celsius degree (C)
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 59 | 64 | 60
Celsius degree (C) | -0.05 (0.307) | -0.07 (0.364) | -0.06 (0.323)

36. Secondary Outcome: Change From Baseline in Vital Signs - Weight
Time Frame: From baseline (day of first dose) to 16 weeks after first dose
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 58 | 63 | 60
Kg | -0.24 (3.690) | 0.18 (2.646) | 0.43 (2.823)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 21 months). Serious Adverse events and other adverse events were assessed from date of first dose to 30 days following date of last dose (up to approximately 13 months).
Description: All participants receiving treatment either only in Part A or in Part A + Part B
Groups:
- Only Part A:Placebo: In Part A, Placebo matching BMS-986165.
- Only Part A:BMS-986165 6 mg QD: In Part A, BMS-986165 6 mg administered QD for 16 weeks.
- Only Part A:BMS-986165 12 mg QD: In Part A, BMS-986165 12 mg administered QD for 16 weeks.
- Part A: Placebo + Part B: Ustekinumab SQ: In Part A, Placebo matching BMS-986165. In Part B, Ustekinumab SQ.
- BMS-986165 6 mg in Part A and Part B: In Part A, BMS-986165 6 mg administered QD for 16 weeks. In Part B, BMS-986165 at 6 mg
- Part A: BMS-986165 6 mg QD - Part B: Ustekinumab SQ: In Part A, BMS-986165 6 mg administered QD for 16 weeks. In Part B, Ustekinumab SQ.
- BMS-986165 12 mg in Part A and Part B: In Part A, BMS-986165 12 mg administered QD for 16 weeks. In Part B, BMS-986165 at 12 mg
- Part A: BMS-986165 12 mg QD - Part B: Ustekinumab SQ: In Part A, BMS-986165 12 mg administered QD for 16 weeks. In Part B, Ustekinumab SQ
Arm/Group | Only Part A:Placebo | Only Part A:BMS-986165 6 mg QD | Only Part A:BMS-986165 12 mg QD | Part A: Placebo + Part B: Ustekinumab SQ | BMS-986165 6 mg in Part A and Part B | Part A: BMS-986165 6 mg QD - Part B: Ustekinumab SQ | BMS-986165 12 mg in Part A and Part B | Part A: BMS-986165 12 mg QD - Part B: Ustekinumab SQ
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/9 | 0/55 | 0/13 | 1/47 | 0/16 | 1/42
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/10 | 0/9 | 0/55 | 1/13 | 3/47 | 0/16 | 4/42
Other Adverse Events (participants affected / at risk) | 6/11 | 7/10 | 7/9 | 34/55 | 13/13 | 30/47 | 11/16 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Only Part A:Placebo (N=11) | Only Part A:BMS-986165 6 mg QD (N=10) | Only Part A:BMS-986165 12 mg QD (N=9) | Part A: Placebo + Part B: Ustekinumab SQ (N=55) | BMS-986165 6 mg in Part A and Part B (N=13) | Part A: BMS-986165 6 mg QD - Part B: Ustekinumab SQ (N=47) | BMS-986165 12 mg in Part A and Part B (N=16) | Part A: BMS-986165 12 mg QD - Part B: Ustekinumab SQ (N=42)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Only Part A:Placebo (N=11) | Only Part A:BMS-986165 6 mg QD (N=10) | Only Part A:BMS-986165 12 mg QD (N=9) | Part A: Placebo + Part B: Ustekinumab SQ (N=55) | BMS-986165 6 mg in Part A and Part B (N=13) | Part A: BMS-986165 6 mg QD - Part B: Ustekinumab SQ (N=47) | BMS-986165 12 mg in Part A and Part B (N=16) | Part A: BMS-986165 12 mg QD - Part B: Ustekinumab SQ (N=42)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 7 | 1 | 6 | 2 | 11
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 2 | 3 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 6 | 2 | 6 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03881059/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT03881059/SAP_001.pdf